CLINICAL TRIAL: NCT04549714
Title: A Prospective,Single Center, Randomized Controlled Trial of Quantitative Ablation of Pulmonary Vein Vestibule in Patients With Paroxysmal Atrial Fibrillation..
Brief Title: Quantitative Ablation of Pulmonary Vein Vestibule in Paroxysmal Atrial Fibrillation.
Acronym: AI-ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuehui Yin (Other)
Responsible Party: Sponsor-Investigator, Yuehui Yin, Director of the Department, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AI-ablation
Record Dates: First submitted 2019-06-07; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation; Arrythmia
Keywords: Atrial Fibrillation; Ablation index; Quantitative Ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients enrolled in the study were randomly assigned to different surgical groups using random envelopes. All study personnel were blind to treatment allocation and had no way of influencing whether a participant would receive high or low AI ablation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High AI in paroxysmal atrial fibrillation (Experimental): In this group,patients with paroxysmal AF will receive pulmonary vein vestibule ablation with high AI value, the AI target value for the front wall and the top wall is 550, and the rear wall and the lower wall are 400.
  Interventions: Procedure: High AI in paroxysmal atrial fibrillation
- Middle AI in paroxysmal atrial fibrillation (Experimental): In this group,patients with paroxysmal AF will receive pulmonary vein vestibule ablation with middle AI value, the AI target value for the front wall and the top wall is 500, and the rear wall and the lower wall are 350.
  Interventions: Procedure: Middle AI in paroxysmal atrial fibrillation
- Low AI in paroxysmal atrial fibrillation (Experimental): In this group,patients with paroxysmal AF will receive pulmonary vein vestibule ablation with low AI value, the AI target value for the front wall and the top wall is 450, and the rear wall and the lower wall are 300.
  Interventions: Procedure: Low AI in paroxysmal atrial fibrillation

INTERVENTIONS:
Procedure: High AI in paroxysmal atrial fibrillation — Patients with paroxysmal AF will receive pulmonary vein vestibule ablation with high AI value, the AI target value for the front wall and the top wall is 550, and the rear wall and the lower wall are 400.
  Arms: High AI in paroxysmal atrial fibrillation
Procedure: Middle AI in paroxysmal atrial fibrillation — Patients with paroxysmal AF will receive pulmonary vein vestibule ablation with middle AI value, the AI target value for the front wall and the top wall is 500, and the rear wall and the lower wall are 350.
  Arms: Middle AI in paroxysmal atrial fibrillation
Procedure: Low AI in paroxysmal atrial fibrillation — Patients with paroxysmal AF will receive pulmonary vein vestibule ablation with low AI value, the AI target value for the front wall and the top wall is 450, and the rear wall and the lower wall are 300.
  Arms: Low AI in paroxysmal atrial fibrillation

SUMMARY:
The purpose of this trial is to explore the optimal AI value for isolating the pulmonary veins and achieving left ventricular apex and mitral isthmus block. Patients with atrial fibrillation who are scheduled to undergo catheter ablation will be randomized to different groups, then every group receive circumferential pulmonary vein isolation with different AI values. The relevant indicators such as the proportion of pulmonary vein single-circle isolation, operation time, the incidence of complications, and the proportion of recurrence of atrial fibrillation and other atrial arrhythmias after 1 year were collected.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial. In this part,a total of 90 patients with paroxysmal atrial fibrillation who are scheduled for catheter ablation were randomly divided into 3 groups, 30 patients in each group. For the first group, the AI target value for the front wall and the top wall is 550, and the rear wall and the lower wall are 400. For the second group, the AI target values for the front wall and the top wall are 500, the rear wall and the lower wall are 350. For the third group, the AI target values for the front wall and top wall are 450, the rear wall and the lower wall are 300. The pressure value at each point is 5-15 g, and the distance between adjacent ablation points is less than 5 mm. The relevant indicators such as single-circle isolation rate of the pulmonary vein, operation time, the left atrial operation time, and the supplemental ablation site are recoded. The incidence of intraoperative and postoperative complications such as stroke, pericardial tamponade and steam pop during ablation are observed. Dynamic electrocardiography is performed during the follow-up period to evaluate the proportion of sinus rhythm within 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female subjects, 18≤age≤80.
2. Receiving or able to tolerate anticoagulant therapy.
3. Diagnosis of atrial fibrillation using an electrocardiogram or a dynamic electrocardiogram
4. The longest duration of atrial fibrillation episode is less than 7 days
5. Patient is compliant and willing to complete clinical follow-up.

Exclusion Criteria:

1. Patients who have previously undergone catheter ablation of atrial fibrillation;
2. Left ventricular ejection fraction <35%;
3. Pregnancy, planned pregnancy or lactating women;
4. Left atrial appendage thrombosis was detected by transesophageal ultrasound or intracardiac ultrasound;
5. Abnormal blood system or liver and kidney function;
6. Combined with severe organic heart disease (including congenital heart disease, valvular heart disease, dilated cardiomyopathy, hypertrophic cardiomyopathy, and patients with myocardial infarction or coronary artery bypass grafting);
7. Patients who are considered unsuitable for inclusion by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of the pulmonary vein single-circle isolation. | Immediately after ablation
  Success rate of the pulmonary vein single-circle isolation.

SECONDARY OUTCOMES:
Total procedure time. | Immediately after ablation
  Time from the start to the end of the ablation procedure
Left atrial operation time. | Immediately after ablation
  Left atrial operation time.
The location and number of supplemental ablation. | Immediately after ablation
  The number and location of the supplemental ablation required for pulmonary vein isolation after single-circle ablation
Intraoperative and postoperative stroke rates. | From the start of procedure to 7 days after ablation
  Intraoperative and postoperative stroke rates.
Intraoperative and postoperative pericardial tamponade rates. | From the start of procedure to 7 days after ablation
  Intraoperative and postoperative pericardial tamponade rates.
Number of steam pop during ablation. | Immediately after ablation
  Number of steam pop during ablation.
the proportion of sinus rhythm within 1 year | 1 year
  Proportion of patients who successfully maintained sinus rhythm within 1 year after ablation.
Recurrence rate of atrial fibrillation | 1 year
  Diagnostic criteria for recurrence of atrial fibrillation: a blank period of 3 months after surgery. After 3 months of ablation surgery, atrial fibrillation/atrial flutter/atrial tachycardia with a duration of more than 30 seconds on the ECG was considered to be a recurrence of atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affilliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Hussein A, Das M, Chaturvedi V, Asfour IK, Daryanani N, Morgan M, Ronayne C, Shaw M, Snowdon R, Gupta D. Prospective use of Ablation Index targets improves clinical outcomes following ablation for atrial fibrillation. J Cardiovasc Electrophysiol. 2017 Sep;28(9):1037-1047. doi: 10.1111/jce.13281. Epub 2017 Jul 26. PMID 28639728
- [Background] Nakagawa H, Ikeda A, Govari A, et al.Prospective study using a new formula incorporating contact force, radiofrequency power and application time (Force-Power-Time Index) for quantifying lesion formation to guide long continuous atrial lesions in the beating canine heart. Circulation2013; 128:A12104.
- [Background] Taghji P, El Haddad M, Phlips T, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Evaluation of a Strategy Aiming to Enclose the Pulmonary Veins With Contiguous and Optimized Radiofrequency Lesions in Paroxysmal Atrial Fibrillation: A Pilot Study. JACC Clin Electrophysiol. 2018 Jan;4(1):99-108. doi: 10.1016/j.jacep.2017.06.023. Epub 2017 Sep 27. PMID 29600792
- [Background] Beinart R, Abbara S, Blum A, Ferencik M, Heist K, Ruskin J, Mansour M. Left atrial wall thickness variability measured by CT scans in patients undergoing pulmonary vein isolation. J Cardiovasc Electrophysiol. 2011 Nov;22(11):1232-6. doi: 10.1111/j.1540-8167.2011.02100.x. Epub 2011 May 26. PMID 21615817